CLINICAL TRIAL: NCT01566760
Title: Open-Label, Single-Dose, Randomized, Crossover Study To Estimate The Effects Of Food On The Pharmacokinetics Of Two Fesoterodine Sustained-Release Beads-In-Capsule Formulations And To Estimate The Relative Bioavailability Of One Or Both Formulations Compared To Commercial Tablet Formulation In Healthy Adult Volunteers
Brief Title: A Study To Estimate The Effects Of Food On Drug Fesoterodine Fumarate And The Pharmacokinetics Of 5-Hydroxymethyl Tolterodine (5-HMT) In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A0221069
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2012-07

CONDITIONS: Urinary Bladder, Overactive
Keywords: food effect; bioavailability; pharmacokinetics; fesoterodine; 5-hydroxymethyl tolterodine; treatment of overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A, Cohort 1 (Experimental)
  Interventions: Drug: fesoterodine fumarate
- Treatment B, Cohort 2 (Experimental)
  Interventions: Drug: fesoterodine fumarate
- Treatment C, Cohort 1 (Experimental)
  Interventions: Drug: fesoterodine fumarate
- Treatment D, Cohort 2 (Experimental)
  Interventions: Drug: fesoterodine fumarate
- Treatment E, Cohort 1 and/or Cohort 2 (Active Comparator)
  Interventions: Drug: fesoterodine fumarate

INTERVENTIONS:
Drug: fesoterodine fumarate — One capsule of 4 mg PF-00695838 Formulation SR1 under fasting conditions, single dose
  Arms: Treatment A, Cohort 1
Drug: fesoterodine fumarate — One capsule of 4 mg PF-00695838 Formulation SR2 under fasting conditions, single dose
  Arms: Treatment B, Cohort 2
Drug: fesoterodine fumarate — One capsule of 4 mg PF-00695838 Formulation SR1 under fed conditions, single dose
  Arms: Treatment C, Cohort 1
Drug: fesoterodine fumarate — One capsule of 4 mg PF-00695838 Formulation SR2 under fed conditions, single dose
  Arms: Treatment D, Cohort 2
Drug: fesoterodine fumarate — one extended-release tablet of commercially available fesoterodine fumarate 4 mg under fasting conditions, single dose
  Arms: Treatment E, Cohort 1 and/or Cohort 2

SUMMARY:
This is an open-label (both the physician and healthy volunteer know which medication will be administered), single-dose, 2-cohort, 3-period study to characterize the pharmacokinetics (process by which drug fesoterodine is absorbed, distributed, metabolized, and eliminated by the body) and the effects of food on the pharmacokinetics of the drug. This study will take place over approximately 8 weeks and will consist of a screening visit to determine eligibility for the study, and 2- or 3-period treatment phase for each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between 21 and 55 years of age(inclusive).

Exclusion Criteria:

* Evidence or history of clinically significant disease.
* Evidence or history of urologic disease (benign prostate hyperplasia, recurrent urinary tract infections, urinary retention, etc.).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve from Time Zero to Extrapolated Infinite Time [AUC(0-inf)] | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, and 48 hours post-dose.
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, and 48 hours post-dose.

SECONDARY OUTCOMES:
Area Under the Curve from Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, and 48 hours post-dose.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, and 48 hours post-dose.
Plasma Decay Half-Life (t1/2) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, and 48 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221069